CLINICAL TRIAL: NCT02722590
Title: Post-Marketing Surveillance of Fycompa in Korean Patients
Brief Title: A Study of Fycompa (Perampanel) in Korean Participants
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M065-505
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Partial-onset seizures; Secondarily generalized seizures; Perampanel; Post marketing surveillance; Primary generalized tonic-clonic seizures; Idiopathic generalized epilepsy
MeSH Terms: conditions — Epilepsy; Epilepsy, Idiopathic Generalized

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants who are prescribed Fycompa (Perampanel) film-coated tablets and oral suspension per approved prescribing information in a normal clinical practice setting will be enrolled and observed prospectively for up to 24 Weeks.

SUMMARY:
The purpose of this post-marketing surveillance is to observe the following items regarding the safety profile of Fycompa (Perampanel) film-coated tablets and oral suspension in normal clinical practice setting: serious adverse event/adverse drug reaction profile, unexpected adverse event/adverse drug reaction profile, already known adverse drug reaction profile, non-serious adverse event profile and other information related to the product's safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with approved indication for Fycompa (Perampanel) in Korea as follows:

   * Monotherapy (film-coated tablets)

     o 4 years and older Partial-onset seizures: therapy for treatment of partial-onset seizures with or without secondarily generalized seizures in participants with epilepsy
   * Adjunctive therapy (film-coated tablets & oral suspension)

     * 4 years and older Partial-onset seizures: therapy for treatment of partial-onset seizures with or without secondarily generalized seizures in participants with epilepsy
     * 7 years and older Primary generalized tonic-clonic seizures: therapy for treatment of primary generalized tonic-clonic seizures in participants with idiopathic generalized epilepsy
2. Participants who have written consent for use of personal and medical information for the study purpose

Exclusion Criteria:

1. Hypersensitivity to the active substance or to any of the excipients of this medicine
2. In case of Fycompa film-coated tablets, Fycompa tablets contains lactose; therefore, participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption should not take this medicine. In case of Fycompa oral suspension, Fycompa suspension contains sorbitol; therefore, participants with rare hereditary problems of fructose intolerance should not take this medicine.
3. Other participants judged to be inadequate to participate in the study by doctor

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female Korean participants who are prescribed with Fycompa (Perampanel) per the approved prescribing information will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3692 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | From the first Fycompa (Perampanel) administration date up to 24 weeks
Number of Participants With Adverse Drug Reactions | From the first Fycompa (Perampanel) administration date up to 24 weeks
Number of Participants With Unexpected Adverse Events | From the first Fycompa (Perampanel) administration date up to 24 weeks
Number of Participants With Serious Adverse Events | From the first Fycompa (Perampanel) administration date up to 24 weeks

SECONDARY OUTCOMES:
Percentage of Participants With Effective Outcome as Measured by Investigator's Clinical Global Impression of Change (CGI-C) Scores | Up to 24 weeks
  The CGI-C score is a clinician's rating scale for assessing Global Improvement of Change. The CGI-C rates improvement by 7 categories: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), very much worse (7). The CGI-C score ranges from 1 to 7, with lower scores indicating improvement. Effective outcome is defined as CGI-C score of: very much improved (1), much improved (2), or minimally improved (3).

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Chungju, Chungcheong-do
  - Wŏnju, Gangwon-do
  - Seongnam, Gyeonggji-do
  - Jinju, Gyeongsang-do
  - Gwangju, Jeolla-do
  - Busan
  - Daegu
  - Daejeon
  - Seoul